CLINICAL TRIAL: NCT02962414
Title: An Open-label, Multi-center Long-term Safety Roll-over Study in Patients With Tuberous Sclerosis Complex (TSC) and Refractory Seizures Who Are Judged by the Investigator to Benefit From Continued Treatment With Everolimus After Completion of Study CRAD001M2304.
Brief Title: Roll-over Study to Collect and Assess Long-term Safety of Everolimus in Patients With TSC and Refractory Seizures Who Have Completed the EXIST-3 Study [CRAD001M2304] and Who Are Benefitting From Continued Treatment
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001M2X02B; 2024-516746-19-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Everolimus; Tuberous sclerosis complex; TSC; Refractory seizure; Roll over study; Long term safety; PASS
MeSH Terms: conditions — Tuberous Sclerosis; Seizures | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- everolimus (Experimental): everolimus, 2mg dispersible tablets
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus, 2mg dispersible tablets
  Other Names: RAD001

SUMMARY:
The purpose of this study is to evaluate the long-term safety in patients with TSC and refractory seizures who are currently receiving everolimus treatment in the Novartis-sponsored EXIST-3 study and who are determined to be benefiting from continued treatment as judged by the investigator at the completion of EXIST-3

DETAILED DESCRIPTION:
This is a multi-center, open label study to evaluate the long term safety of everolimus in patients with TSC and refractory seizures currently being treated in the Novartis-sponsored study EXIST-3 study and are judged by their parent study investigator as benefiting from the current study treatment. The study is expected to remain open for approximately 10 years (or until 31-Dec-2022 in the UK) from First Patient First Visit (FPFV).

Patients will continue to be treated in this study until they are no longer benefiting from their everolimus treatment as judged by the Investigator or until one of the protocol defined discontinuation criteria is met or everolimus becomes commercially available according to local regulations.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is currently enrolled in the Novartis-sponsored EXIST-3 study, receiving everolimus, and has fulfilled all its requirements
* Patient is currently benefiting from treatment with everolimus, as determined by the Investigator.
* Patient has demonstrated compliance, as assessed by the Investigator,with the parent study protocol requirements.
* Patient is willing and able to comply with scheduled visits and treatment plans.
* Written informed consent/adolescent assent obtained prior to enrolling into the roll-over study.

Key Exclusion Criteria:

* Patient has been permanently discontinued from everolimus study treatment in EXIST-3 study
* Everolimus is approved for patients with TSC and refractory seizures and is reimbursed in the local country.
* Patients who are receiving everolimus in combination with unapproved or experimental treatments for seizure control Anti-epileptic drug (AEDs) are allowed for the purpose of seizure control.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2027-08-04 (Estimated); Study Completion 2027-08-13 (Estimated)

PRIMARY OUTCOMES:
Occurances of adverse events and serious adverse events | Day 1 up to approximately 10 years
  The patients will be followed continuously for tolerability (i.e adverse events, serious adverse events)

SECONDARY OUTCOMES:
Percentage of patients with clinical benefit | Day 1 up to approximately 10 years, assessed every 12 weeks,
  At every quarterly visit (every 12 weeks ± 2 weeks), the Investigator is required to confirm that the patients continue to have clinical benefit as per Investigator's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (14):
  - TGen APNNA, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UCSF Benioff Children s Hospital, Oakland, California
  - Rady Children s Hospital, San Diego, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Connecticut Childrens Medical Cntr, Hartford, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Atlantic Health Systems, Morristown, New Jersey
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Scottish Rite Hos for Child, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- Novartis Investigative Site, Cali, Valle del Cauca Department, Colombia
- France (5):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Strasbourg
- Novartis Investigative Site, Budapest, Hungary
- Italy (5):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
- Japan (4):
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Novartis Investigative Site, Warsaw, Poland
- Russia (3):
  - Novartis Investigative Site, Samara, Samara Oblast
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Voronezh
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Donostia / San Sebastian, Gipuzkoa
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Ankara, Yenimahalle
- United Kingdom (7):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Buckinghamshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com